CLINICAL TRIAL: NCT02459808
Title: Gastrointestinal Transit Time in Patients With Guillain-Barré Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Inclusion according to criteria was not practical in our setting.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: GBSTransitTimeAarhus
Record Dates: First submitted 2015-05-18; First posted 2015-06-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2015-04

CONDITIONS: Guillain-Barre Syndrome; Constipation
MeSH Terms: conditions — Guillain-Barre Syndrome; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GBS Patients: Patients with Guillain-Barré syndrome

SUMMARY:
Constipation is a common condition among patients with Guillain-Barré Syndrome. It is believed, that the constipation is caused by autonomic neuropathy. However, the severity of the constipation, and its relation to autonomic function have not previously been studied.

ELIGIBILITY:
Inclusion Criteria:

* Guillain-Barré Syndrome
* Ability to swallow the capsules used to assess GITT
* Ability to give meaningful informed consent to participate in the study

Exclusion Criteria:

* Major abdominal disorders
* Severe acute comorbidity
* Known cancer
* Pregnancy
* Other known neurological disorder
* Use of laxatives one week before inclusion. (Patients will be excluded if medication with laxatives is started during the one week GITT measurement)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Aarhus University Hospital, admitted with Guillain-Barré syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal transit time (GITT) [in days] | The measurement takes one week to perform. The investigators aim to start the measurement within one week after diagnosis.

SECONDARY OUTCOMES:
Association between heart rate variability (HRV) and GITT | The first HRV measurement is performed within one week after diagnosis. The second is performed 7 days after the first.
  Linear regression with GITT as dependent variable, and high frequency power spectral density analysis of the heart rate (HF) as the independent variable. The mean HF of the first and second HRV measurement is used for this regression.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Dr. med. PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark